CLINICAL TRIAL: NCT02235636
Title: Da Vinci Robot Compared to Laparoscopic Suturing for Closure of Gastric Incision Among Novice: a Randomized Cross Over Trial
Brief Title: A Randomized Cross-over Trial of Comparison Between Robotic and Laparoscopic Suturing for Gastric Defect by Novices
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan Chiu, Professor, Chinese University of Hong Kong
Other Study IDs: 098-12
Record Dates: First submitted 2014-09-04; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Surgical Suturing for Closure of Gastrotomy; Laparoscopic Suturing; Robotic Surgical Suturing

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laparoscopic group
- Robotic group

SUMMARY:
To compare the performance of surgical suturing using Da Vinci Robotic Surgical System and conventional Laparoscopic surgical suturing among novice

DETAILED DESCRIPTION:
Background Da Vinci® Robotic Surgical System (DVRSS) has been widely applied to perform complex minimally invasive surgical procedures across different specialties. This study aimed to investigate the impact of DVRSS on surgical proficiencies among inexperience novice surgeons and compared to conventional laparoscopic surgery.

Methods Twenty medical students (n=20) without surgical experience were enrolled. After a constructive training for basic surgical techniques, participants were randomly allocated into DVR or laparoscopy group. Participants were asked to close five cases (also named five tasks) of a 2cm long incision on pig stomach by using DVR or laparoscopy. Surgical time, successful closure rate and pneumatic bursting pressure of gastric incision withstanding were recorded. In addition, participant performance and workload were quantified by using performance score, scales of Global Rating Scale Assessment (GSA) and NASA-Task Load Index (NASATLI).

ELIGIBILITY:
Inclusion Criteria:

* Medical Students with no prior surgical experience

Exclusion Criteria:

* Surgeons
* Age < 16 or > 60
* Disability and not able to control the Da Vinci Robot through the console

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Medical students with no prior experience in surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Task performance | 1 day
  The performance of participants for each task would be assessed by objective scoring scale basing on the task completion time, plus well-defined errors during suturing and tying knot.

SECONDARY OUTCOMES:
Rate of success in closure of gastrotomy | 1 day
  The success in closure of the standardized gastrotomy was defined as followings: (1) The gastrotomy must be closed with 20 minutes using a 10 cm-long suture with intracorporeal knots tying; (2) Sutures should not be broken during the experiment.
Pneumatic bursting pressure for gastric incision | 1 day
  The efficiency of the two groups in using DVRSS and laparoscopic suturing for closure of gastrotomy was assessed by the maximal pneumatic bursting pressure that the suture line could withstand.
Assessment of participant workload | 1 day
  Participant workload was assessed by using National Aeronautics and Space Administration-task load index scale (NASATLX) after completion of each task. The scale focused on six domains, including mental, physical and temporal demand, as well as performance, effort and frustration.

CONTACTS AND LOCATIONS:
Overall Officials: Philip W Chiu, MD, Principal Investigator — Department of Surgery, The Chinese University of Hong Kong
Locations (1):
- CUHK Jockey Club Minimally Invasive Surgical Skills Center, Hong Kong SAR, China